CLINICAL TRIAL: NCT00113672
Title: Multiple Behavior Change in Diet and Activity
Brief Title: Make Better Choices Study
Acronym: MBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bonnie Spring, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 182; R01HL075451 (NIH)
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Increase healthy eating and increase healthy activity
  Interventions: Behavioral: Increase healthy activity and increase healthy eating
- B (Experimental): Increase healthy eating and decrease unhealthy activity
  Interventions: Behavioral: Decrease unhealthy activity and increase healthy eating
- C (Experimental): Decrease unhealthy eating and increase healthy activity
  Interventions: Behavioral: Increase physical activity and decrease unhealthy eating
- D (Experimental): Decrease unhealthy activity and decrease unhealthy eating
  Interventions: Behavioral: Decrease sedentary activity and decrease unhealthy eating

INTERVENTIONS:
Behavioral: Increase healthy activity and increase healthy eating — Increase participants to 60 minutes of activity per day and 5 fruits and vegetables per day over a 3 week prescription phase
  Arms: A
Behavioral: Decrease unhealthy activity and increase healthy eating — Decrease sedentary activity by 90 minutes per day and increase fruits and vegetables to 5 servings per day over the course of a 3 week prescription phase
  Arms: B
Behavioral: Increase physical activity and decrease unhealthy eating — Increase physical activity up to 60 minutes per day and decrease saturated fat to an average of 8% per day over the course of a 3 week prescription phase
  Arms: C
Behavioral: Decrease sedentary activity and decrease unhealthy eating — Decrease sedentary activity by 90 minutes per day and decrease saturated fat to and average of 8% per day over the course of a 3 week prescription phase
  Arms: D

SUMMARY:
The purpose of this study is to examine the impact of diet and exercise on an individual's health.

DETAILED DESCRIPTION:
BACKGROUND:

The majority of adult Americans consume a high saturated fat diet, have a low fruit and vegetable (F/V) intake, and lead a sedentary lifestyle. This unhealthy lifestyle heightens their risk for cardiovascular disease and cancer. Improving diet and activity can reduce risk, but the best prescription to promote a healthier diet and a more active lifestyle remains unknown. This study will randomly assign participants to 4 groups, which will include all combinations of increasing healthy eating and activity and decreasing unhealthy eating and activity. The Familiarity Hypothesis predicts that the most familiar dieting prescription (decrease fat, increase physical activity) will maximize healthy behavior change. The Optimal Substitution Hypothesis, based on Behavioral Economic Theory, predicts that increasing F/V intake while decreasing sedentary behavior will surpass alternative methods by maximizing behavioral substitution of healthful eating and activity for unhealthful eating and activity. The Low Inhibitory Demand Hypothesis, based on Self-Control Theory, predicts that increasing F/Vs while increasing physical activity will be most successful because this prescription places the fewest demands on self-control resources.

DESIGN NARRATIVE:

The study will randomize 200 sedentary community-dwelling adults with a suboptimal diet to 1 of 4 groups including: 1) increase healthy eating and activity; 2) decrease unhealthy eating and activity; 3) increase healthy eating and decrease unhealthy activity; and 4) decrease unhealthy eating and increase healthy physical activity. Subjects will self-monitor diet, physical activity, and mood via PDAs during a 2-week baseline period, a 3-week prescription period (when payment is contingent upon changing eating and activity simultaneously to targeted standards), and a 4-month maintenance period. Targeted and collateral diet and activity changes will be measured by self report, accelerometer, and grocery receipts. Bogus pipeline urinary testing will encourage adherence. Laboratory testing will measure behavioral choices, craving, and attentional allocation to restricted foods and activities in a permissive context in order to shed light on behavioral and psychological processes that mediate healthy lifestyle change. Findings will help to fill an important gap in clinical knowledge about how to optimize healthy simultaneous change in diet and activity among adults.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary community dwelling adults with a suboptimal diet
* Motivated to make changes in diet and activity level

Exclusion Criteria:

* Few exclusion criteria will be implemented in order to enhance generalizability
* For safety, participants with unstable medical conditions (uncontrolled hypertension, diabetes, recent myocardial infarction) will be excluded. Those with stable medical conditions will require physician approval to participate but will not be excluded because the prescribed changes in diet and activity match healthy, attainable guidelines for all Americans.
* Cannot read the study questionnaires
* Committed to following an incompatible dietary regimen
* Pregnant, trying to get pregnant, or breastfeeding
* People with anorexia, bulimia, or report active suicidal ideation will not be enrolled because they might practice overly severe dietary restrictions
* Binge eating disorder
* Current substance abuse or dependence, other than nicotine dependence will be excluded because of concern about their ability to maintain accurate records of intake and activity. Smokers will be accepted and during recreational laboratory sessions will be able to smoke cigarettes in an adjoining room that is used as a smoking laboratory.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2004-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Daily diet and activity (measured at Week 1 and 3, and Month 1, 2, 3, 4, 5, and 6) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Welch WA, Groth CP, Phillips SM, Spring B, Siddique J. Comparing Accelerometer and Self-Reported Treatment Effects in a Technology-Supported Physical Activity Intervention. Health Educ Behav. 2021 Feb;48(1):34-41. doi: 10.1177/1090198120971194. Epub 2020 Nov 13. PMID 33185131
- [Derived] Spring B, Schneider K, McFadden HG, Vaughn J, Kozak AT, Smith M, Moller AC, Epstein L, Russell SW, DeMott A, Hedeker D. Make Better Choices (MBC): study design of a randomized controlled trial testing optimal technology-supported change in multiple diet and physical activity risk behaviors. BMC Public Health. 2010 Sep 29;10:586. doi: 10.1186/1471-2458-10-586. PMID 20920275